CLINICAL TRIAL: NCT00805558
Title: Comparison of Moxifloxacin With Ciprofloxacin/Metronidazole as Adjunctive Therapy to Mechanical Treatment of Patients With Chronic Periodontitis
Brief Title: Comparison of Moxifloxacin With Ciprofloxacin/Metronidazole on Patients With Chronic Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Facultad Nacional de Salud Publica (Other)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Carlos Martín Ardila Medina, Grupo Epidemiologia Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARD-0001-CM; CBEIH-SIU 08-44-203
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Periodontitis
Keywords: Chronic Periodontitis; antibiotics
MeSH Terms: conditions — Chronic Periodontitis | interventions — Moxifloxacin; Ciprofloxacin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxifloxacin (Experimental): Scaling and root planing plus 400 mg moxifloxacin once daily for 7 days.
  Interventions: Drug: moxifloxacin
- Ciprofloxacin plus metronidazole (Active Comparator): Scaling and root planing plus ciprofloxacin 1000 mg once daily for 7 days and metronidazole 500 mg twice daily for 7 days
  Interventions: Drug: Ciprofloxacin plus metronidazole

INTERVENTIONS:
Drug: moxifloxacin — 400 mg moxifloxacin once daily for 7 days
  Other Names: Moxifloxacin hydrochloride
  Arms: Moxifloxacin
Drug: Ciprofloxacin plus metronidazole — Ciprofloxacin 1000 mg once daily for 7 days; Metronidazole 500 mg twice daily for 7 days
  Other Names: ciprofloxacino; metronidazole benzoato
  Arms: Ciprofloxacin plus metronidazole

SUMMARY:
The purpose of this study is to assess the clinical and microbiological effectiveness of the moxifloxacin compared with the combination ciprofloxacin - metronidazole, when used as adjunctive therapy to scaling and root planning for the treatment of advanced chronic periodontitis.

DETAILED DESCRIPTION:
Periodontitis is an endemic inflammatory disease caused by a mixed bacterial biofilm infection that is followed by destruction of tooth supporting tissues. Standard of care consists of lifelong mechanical removal of the biofilm. However, outcome is variable. According to recent EFP and AAP reviews, adjunctive antimicrobial therapy may be beneficial.However, bearing in mind that Colombia has reported the frequent presence of Enterobacteriaceae (Klebsiella and Enterobacter) in subgingival plaque of patients with chronic periodontitis, the response to treatment may be different.The enteric have shown resistance to amoxicillin, amoxicillin / clavulanate, metronidazole and tetracycline in studies conducted in the United States, Norway, Brazil and Colombia.Although the combination ciprofloxacin metronidazole has been recommended in the dental literature are not known publications that demonstrate its effectiveness against periodontopathogens and enteric present in subgingival plaque of subjects with chronic periodontitis.On the other hand, some in vitro studies have demonstrated the effectiveness of moxifloxacin against periodontopathogens, but was not aware of any clinical trials or in vitro studies on antibiotic resistance and susceptibility to enteric isolated subgingival plaque of patients with chronic periodontitis in which employs moxifloxacin.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and up
* clinical and radiographic signs of severe (CAL 5 mm or more) chronic periodontitis.
* at least 20 natural teeth in situ
* pocket probing depths (PPDs) of ≥ 5 mm at a minimum of eight tooth sites
* willingness to participate and to be available at all times required for participation
* over 30% of the teeth present must have a PPDs)≥ 4 mm and insertion loss ≥ 5 mm evaluated by an experienced periodontist
* informed consent signed by the patient

Exclusion Criteria:

* if they (or parents or siblings) show confirmed or assumed allergies or hyper-sensitive skin reactions against moxifloxacin, ciprofloxacin (or other quinolones as listed in the "summary of product characteristics, Version Juli 2005"), metronidazole (or other 5-nitroimidazoles and ingredients of Flagyl® 400mg as listed in the "summary of product characteristics, Version Juli 2007"), systemic diseases or conditions as listed in the above mentioned "summary of product characteristics"
* subjects who have undergone antibiotic therapy three months before the start of the study under interrogation
* have Down's syndrome
* known AIDS/HIV
* regularly take systemic medication affecting the periodontal conditions, e.g. phenytoin, nifedipine, and/or steroid drugs
* professional periodontal therapy during 6 months prior to baseline
* require antibiotic treatment for dental appointments
* are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Probing Depth | six months period (two measurements)

SECONDARY OUTCOMES:
Subjective perception of treatment outcome, attachment gain,bleeding on probing, and full mouth plaque score. | six months
Microbial colonization dynamic | six months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Ardila, DDS Cand PhD, Principal Investigator — Grupo Epidemiologia Universidad de Antioquia
Locations (1):
- Faculta Nacional de Salud Publica Universidad de Antioquia, Medellín, Antioquia, Colombia

REFERENCES:
- [Result] Ardila CM, Fernandez N, Guzman IC. Antimicrobial susceptibility of moxifloxacin against gram-negative enteric rods from colombian patients with chronic periodontitis. J Periodontol. 2010 Feb;81(2):292-9. doi: 10.1902/jop.2009.090464. PMID 20151809
- [Result] Ardila CM, Lopez MA, Guzman IC. High resistance against clindamycin, metronidazole and amoxicillin in Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans isolates of periodontal disease. Med Oral Patol Oral Cir Bucal. 2010 Nov 1;15(6):e947-51. PMID 20383102
- [Derived] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289
- See also: Clinical trial of moxifloxacin in chronic periodontitis — http://www.udea.edu.co